CLINICAL TRIAL: NCT05076448
Title: Evaluation of the Efficacy and Safety of Surgical and Endovascular Interventions on the Pelvic Veins in Pelvic Venous Disorders
Brief Title: The Efficacy and Safety of Interventions on the Pelvic Veins in Pelvic Venous Disorders
Acronym: ESIPV
Status: Completed | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Sergey Gavrilov, MD, PhD, Professor, Pirogov Russian National Research Medical University
Other Study IDs: 012012548111
Record Dates: First submitted 2021-09-20; First posted 2021-10-13 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Pelvic Venous Disorders; Pelvic Congestive Syndrome; May-Thurner Syndrome
Keywords: Pelvic Venous Disorders; Pelvic Pain; Gonadal Veins Resection; Gonadal veins Embolization; Iliac vein stenting; Complications of pelvic vein interventions
MeSH Terms: conditions — May-Thurner Syndrome; Pelvic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Gonadal veins resection This group includes patients who underwent open retroperitoneal resection of the gonadal veins, endoscopic transperitoneal and retroperitoneal resection of the gonadal veins.
  Interventions: Procedure: Gonadal veins resection
- 2: Gonadal veins embolozation This group includes patients who underwent embolization of the gonadal veins with coils.
  Interventions: Procedure: Gonadal vein embolization with coils
- 3: Stenting of the common iliac vein with or without gonadal veins embolization This group includes patients who underwent isolated iliac vein stenting or iliac vein stenting combined with gonadal vein embolization.
  Interventions: Procedure: Endovascular stenting of the common iliac vein (CIV)

INTERVENTIONS:
Procedure: Gonadal veins resection — Gonadal veins resection (GVR) was performed open, transperitoneal and retroperitoneal endoscopic methods under general anesthesia.
  Open GVR was performed in the Trendelenburg position, on the back with the operating table rotating 30° The retroperitoneal approach was employed in the left and/or right iliac region. The GV was mobilized for 10-12 cm and the vein was resected..
  Transperitoneal GVR was performed with 3 ports were placed: one 10-mm port in the umbilical region, one 5-mm port in the left or right iliac region, and one 5-mm port 5 cm below the umbilicus. The GV was mobilized over a length of 10-12 cm and the vessel was resected.
  Retroperitoneal GVR was performed with the patient in a lateral position and in the reverse Trendelenburg position. A 10-mm camera port was installed in the lumbar region between the posterior superior iliac spine and the lower edge of the XII rib. The GV was mobilized over a length of 10-12 cm and the vessel was resected.
  Groups: 1
Procedure: Gonadal vein embolization with coils — Procedure was performed under local anesthesia with 5.0-10.0 mL of 0.5% lidocaine solution with a patient under intravenous sedation. For the left GV embolization, the transfemoral approach was used, while for the right or both GV embolization, the transjugular approach was used. The vein puncture was performed under ultrasound guidance. The 5F multipurpose angiographic catheters (Cordis; USA), standard 'moving core' J .035" guidewire, and an angled hydrophilic guidewire (Radiofocus; Terumo Corp., Japan) were used. For the GV occlusion, the pushable 0.035" standard stainless steel coils (Gianturco; William Cook, Bjæverskov, Denmark) and 0.035" coils made of Inconel with interwoven long collagen fibrils (MReye; Cook Medical Inc., Bloomington, USA) were used. The diameter of coils was 8-12 mm, and the length was 10-20 cm.
  Groups: 2
Procedure: Endovascular stenting of the common iliac vein (CIV) — After providing local anesthesia, the left common femoral vein was punctured, a 0.035" guidewire was inserted into the inferior vena cava (IVC), and then a 10F introducer was installed. A balloon catheter was introduced over the guidewire in the left CIV (XXL balloon, Boston Scientific, diameter 14-18, length 40-60 mm), and double balloon dilation of the vessel was performed with a pressure of 6-8 atm. Then, a delivery system was advanced to the area of stenosis in the left CIV, and stent was deployed at the level of confluence of the left CIV and inferior vena cava (IVC) or with a protrusion in the IVC of no more than 1 cm. For better fixation of stent in the venous lumen and prevention of its displacements and migration, a balloon post-dilatation of the stented vessel was performed. In case of residual stenosis, the balloon angioplasty was performed.
  Groups: 3

SUMMARY:
This study includes a retrospective and prospective study will enroll patients with pelvic venous disorders who have undergone pelvic vein surgery and endovascular interventions. Three groups of patients will be formed. The first will include patients who underwent open retroperitoneal resection of the gonadal veins and endoscopic trans- and retroperitoneal resection of the gonadal veins. The second group will include patients who underwent embolization of the gonadal veins with coils, the third - patients who underwent stenting of the common iliac veins, or stenting of the iliac veins in combination with embolization of the gonadic veins with coils. Evaluation of the effectiveness and safety of interventions on the pelvic veins will be carried out by assessing the effect of the intervention on pelvic pain, morphological and functional state of the pelvic veins. The assessment of the safety of interventions on the pelvic veins will be carried out by assessing the severity of post-procedural pain, the frequency of complications of operations on the pelvic veins, and complications of anesthesia. In addition, the duration of pelvic vein interventions will be compared with the length of time the patient is in hospital. Based on the data obtained, an algorithm will be proposed for determining the choice of the method of interventions on the pelvic veins in patients with pelvic venous disorders.

DETAILED DESCRIPTION:
This study includes a retrospective and prospective study and will include patients with pelvic venous disorders (ovarian venous insufficiency, compression stenosis of the left or right common iliac vein) who underwent surgical and endovascular interventions on the pelvic veins during 2000-2022. The database of the local system "Interin" of the First City Hospital of Moscow (Russia) will be used, into which all information about patients with pelvic venous diseases during 2000-2021 was entered.

In this study, the pelvic veins included the gonadal, parametric, uterine, common, external and internal iliac veins.

Indications for intervention on the gonadal veins are symptoms and signs of pelvic venous disorder (pelvic pain, dyspareunia, heaviness in the hypogastric region, vulvar varicose veins) in combination with the expansion of the gonadal veins of more than 5 mm and reflux in them for more than 1 s.

The indication for intervention on the left / right common iliac vein is the presence of compression stenosis of these veins of more than 50% in combination with symptoms and signs of pelvic venous disease.

Three groups of patients will be formed. The first will include patients with ovarian venous insufficiency, dilation of the gonadal veins of more than 10 mm and reflux along them for more than 1 s, who underwent open retroperitoneal resection and endoscopic trans- and retroperitoneal resection of the gonadal veins.

The second group will include patients with ovarian venous insufficiency, dilatation of the gonadal veins less than 10 mm and pelvic venous reflux for more than 1 s, who have undergone embolization of the gonadal veins with coils.

The third will include patients with a combination of May-Thurner-Cockett syndrome and pelvic congestion syndrome who have stenting of the common iliac veins, or stenting of the iliac veins in combination with embolization of the gonadal veins with coils.

Evaluation of the effectiveness and safety of interventions on the pelvic veins will be carried out by assessing the effect of the intervention on pelvic pain, morphological and functional state of the pelvic veins. A visual analogue scale will be used to assess the dynamics of pelvic pain after gonadal and iliac vein interventions.

The assessment of the morphological and functional state will be carried out using the results of transabdominal and transvaginal duplex ultrasound (diameter of the pelvic veins, linear blood flow velocity through them, the presence of reflux in these veins and its duration).

The assessment of the safety of interventions on the pelvic veins will be carried out by assessing the severity of post-procedural pain, the frequency of complications of operations on the pelvic veins, and complications of anesthesia.

Postoperative / Postprocedural pain was assessed using a visual analogue scale.

Complications of gonadal and iliac vein interventions were assessed within 1-30 days after surgery. Complications of gonadal vein resection included:

1. Wound infectious complications;
2. Thrombosis of non-targeted pelvic veins (parametric, uterine, internal iliac veins);
3. Bleeding with the formation of a retroperitoneal hematoma after surgery;
4. Massive bleeding during surgery;
5. Intestinal paresis (ileus).

Complications of gonadal vein embolization with coils included:

1. Hematoma / bleeding at the access point;
2. Thrombosis of non-targeted pelvic veins (parametric, uterine, internal iliac veins);
3. Postembolization syndrome;
4. Protrusion of spirals;
5. Migration of spirals;
6. Allergic reactions to contrast agent or nickel.

Complications of stenting of the common iliac vein included:

1. Hematoma / bleeding at the access point;
2. Stent thrombosis;
3. Migration of the stent;
4. Perforation of the iliac veins or inferior vena cava. In addition, the duration of pelvic vein interventions will be compared with the length of time the patient is in hospital.

ased on this study of data, objective information will be obtained on the effectiveness and safety of interventions on the gonadal and iliac veins, and an algorithm will be proposed for determining the choice of the method of interventions on the pelvic veins in patients with pelvic venous disorders.

ELIGIBILITY:
Inclusion Criteria:

* the presence of pelvic venous disorder symptoms and signs (chronic pelvic pain, dyspareunia, discomfort/heaviness in the hypogastrium);
* reflux in the gonadal, parametrial, uterine veins, according to duplex ultrasound scanning and ovarian venography or multislice computed venography (MSCV);
* narrowing of the lumen of the left CIV greater than 50% with imaging of collateral veins by the radiological contrast studies

Exclusion Criteria:

* combined surgery on the veins and pelvic organs; comorbidities with СРР

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: This single-center retrospective cohort study included female patients with pelvic venous disorders caused by valvular incompetence of the gonadal, parametrial and uterine veins and May-Thurner syndrome, who were treated at the Savelyev University Surgical Clinic of the Pirogov Russian National Research Medical University in the period from 2000 to 2021.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-11 (Actual)

PRIMARY OUTCOMES:
Change in the severity of pelvic pain | At baseline and 12 months after pelvic vein intervention.
  The visual analogue scale is a line 10 cm long. Each centimeter corresponds to 1 point: 0 points - no pain, 10 points - maximum pain. Higher scores on the scale correspond to poorer results.

SECONDARY OUTCOMES:
Change in the diameter of the pelvic veins | At baseline and 12 months after pelvic vein intervention.
  The diameter of the pelvic veins was measured using duplex ultrasound.
Change in the duration of pelvic venous reflux | At baseline and 12 months after pelvic vein intervention.
  Pelvic venous reflux was measured using duplex ultrasound. Reflux duration of more than 1 s was considered pathological.
Postprocedural pain | 1 day, 5 days, 1 and 12 months after the intervention on the pelvic veins.
  The visual analogue scale is a line 10 cm long. Each centimeter corresponds to 1 point: 0 points - no pain, 10 points - maximum pain. Higher scores on the scale correspond to poorer results.
Pelvic vein thrombosis | 1 and 5 days after the intervention on the pelvic veins
  Pelvic vein thrombosis was detected using duplex ultrasound.

OTHER OUTCOMES:
Complications of anesthesia | 1 and 5 days after the intervention on the pelvic veins
  Hematoma, vascular damage, pulmonary complications.
Wound infectious complications | 5 days after the intervention on the pelvic veins
  It was assessed visually, on the basis of examination and palpation of the puncture point of the main vein or postoperative wounds.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia V Koroleva, PhD, Study Director — Pirogov Russian National Research Medical University
Locations (1):
- Department of Faculty Surgery №1, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lakhanpal G, Kennedy R, Lakhanpal S, Sulakvelidze L, Pappas PJ. Pelvic venous insufficiency secondary to iliac vein stenosis and ovarian vein reflux treated with iliac vein stenting alone. J Vasc Surg Venous Lymphat Disord. 2021 Sep;9(5):1193-1198. doi: 10.1016/j.jvsv.2021.03.006. Epub 2021 Mar 18. PMID 33746048
- [Result] Maratto S, Khilnani NM, Winokur RS. Clinical Presentation, Patient Assessment, Anatomy, Pathophysiology, and Imaging of Pelvic Venous Disease. Semin Intervent Radiol. 2021 Jun;38(2):233-238. doi: 10.1055/s-0041-1729745. Epub 2021 Jun 3. PMID 34108811
- [Result] Meissner MH, Khilnani NM, Labropoulos N, Gasparis AP, Gibson K, Greiner M, Learman LA, Atashroo D, Lurie F, Passman MA, Basile A, Lazarshvilli Z, Lohr J, Kim MD, Nicolini PH, Pabon-Ramos WM, Rosenblatt M. The Symptoms-Varices-Pathophysiology classification of pelvic venous disorders: A report of the American Vein & Lymphatic Society International Working Group on Pelvic Venous Disorders. J Vasc Surg Venous Lymphat Disord. 2021 May;9(3):568-584. doi: 10.1016/j.jvsv.2020.12.084. Epub 2021 Jan 30. PMID 33529720
- [Result] Possover M, Khazali S, Fazel A. Pelvic congestion syndrome and May-Thurner syndrome as causes for chronic pelvic pain syndrome: neuropelveological diagnosis and corresponding therapeutic options. Facts Views Vis Obgyn. 2021 Jun;13(2):141-148. doi: 10.52054/FVVO.13.2.019. PMID 34184843

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT05076448/Prot_SAP_000.pdf